CLINICAL TRIAL: NCT05653635
Title: Contribution From PET-DOPA in Glioblastoma Re-irradiation - A Randomized Phase II Study
Acronym: ReciDOPA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Paul Strauss (Other)
Collaborators: Centre Georges François Leclerc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-011
Record Dates: First submitted 2022-11-28; First posted 2022-12-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Simultaneous Integrated Boost
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simultaneous-integrated boost with Intensity-modulated radiation therapy (IMRT) (Experimental): * Planning Target Volume (PTV) 37,5 Gray (Gy): 37,5 Gy in 6 fractions of 6,25 Gy at the rate of one fraction each 2 days
  * Prescription isodose line (PIL) at 80%, corresponding to 30 Gy as total dose, or 5 Gy per fraction
  * PTV SIB 45 Gy: 45,0 Gy in 6 fractions of 7,50 Gy at the rate of one fraction each 2 days
  * PIL at 80% corresponding to 36 Gy as total dose, or 6 Gy per fraction
  Interventions: Radiation: Simultaneous-integrated boost with IMRT
- Standard IMRT (No Intervention): * PTV 37,5 Gy: 37,5 Gy in 6 fractions of 6,25 Gy at the rate of one fraction each 2 days
  * PIL at 80%, corresponding to 30 Gy as total dose, or 5 Gy per fraction
  * No SIB

INTERVENTIONS:
Radiation: Simultaneous-integrated boost with IMRT — Simultaneous-integrated boost guided by FDOPA-PET
  Arms: Simultaneous-integrated boost with Intensity-modulated radiation therapy (IMRT)

SUMMARY:
ReciDOPA is a phase II, single-stage randomized, multicenter, prospective trial assessing the efficacy of an irradiation protocol based on Intensity-modulated radiation therapy with simultaneous-integrated boost guided by FDOPA-PET in patient with recurrent glioblastoma.

DETAILED DESCRIPTION:
Glioblastoma (GBM) is the most common cerebral tumor in adults. Despite well-conducted treatments including surgery, chemo-radiotherapy and chemotherapy according to the European Organisation for Research and Treatment of Cancer (EORTC) and National Cancer Institute of Canada Clinical Trials Group (NCIC) protocol, recurrences remain unavoidable within approximately 6 months and the overall survival rate of patients at 5 years is inferior to 10%.

In case of recurrence, a second surgery, radiotherapy under stereotaxic conditions, bevacizumab or other innovative techniques have been proposed. However, they are not yet considered as reference treatments, due to the absence of therapeutic trials definitively proving their efficacy.

Evaluation of GBM progression is based on MRI, corticosteroid intake and clinical status.However, positron emission tomography (PET) is an extremely relevant examination for differentiating between true progression and pseudo-progression. Indeed, an increase in the transfer of amino acids in 18 F-dihydroxyphenylalanine (FDOPA)-PET strongly suggests a recurrence. A local treatment can then be proposed by favoring surgery or, as an option, radiotherapy under stereotactic conditions. However, this treatment, even if it is well tolerated, has an efficacy which could be improved.

Often proposed option to improve efficacy of this radiation technic consists in increasing the dose of irradiation. This dose increase is often limited by the tolerance of nearby healthy tissue. It could however be possible with coupled techniques of intensity modulation and stereotaxy within the framework of an integrated boost (Simultaneous Integrated Boost - SIB). At each radiation session, the dose delivered to the tumor volume would be increased in the metabolic volume (BTV) detected by FDOPA-PET.

The objective of this study is to evaluate, in patients with recurrent glioblastoma, the efficacy of a dose increase using an SIB in a volume delineated with FDOPA-PET.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Glioblastoma, World Health Organization (WHO) grade IV, histologically proven
* Performance status 0, 1 or 2
* Neurological status ≥ 2
* Past irradiation in previsional re-irradiated site or in the vicinity (5 to 7 cm)
* Radiological proven recurrence according to 1 and 2 criteria, Wen et al
* Remaining node after partial surgery post-recurrence
* 1 to 3 recurrence site(s) < 35 mm in wide axis and separated by at least 5 mm
* Volume of each lesion < 35 mL
* Distance between recurrence node(s) and optic nerves (left and right), chiasma and/or cerebral trunk > 10 mm

Exclusion Criteria:

* Patient with contraindication to MRI or PET
* Glioblastomatose
* Pregnancy or breastfeeding
* Patient that do not understand French
* Patient without affiliation to the national or local social security
* Patients not able to comply to the protocol assessments for geographic, social or psychological reasons
* Minor or patients placed under guardianship or supervision
* Patients deprived of liberty
* Patients placed under judicial protection
* Patients that are not able to express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of simultaneous-integrated boost with IMRT guided by FDOPA PET on Recurrence free survival in patient with recurrent glioblastoma | up to 24 months
  Recurrence free survival: interval between the date of inclusion in the trial until the date of recurrence of irradiated site (or one of the irradiated sites, in case of multiple irradiation)

SECONDARY OUTCOMES:
Percentage of recurrence of irradiated sites | up to 24 months
  Number of sites with recurrence over the number of irradiated sites
Characterization of recurrence sites: classified either as distant, marginal or in-field | up to 24 months
  Recurrence will be described according to their localisation by comparing images at recurrence with the images used for dosimetry. A recurrence will be defined as " distant" is it appears outside of 80% isodose, as "marginal" if it cuts 80% isodose and as "in-field" if it is completely located in 80% isodose. The 80% isodose is the reference isodose used for radiation therapy prescription.
Percentage of Recurrence free survival at 6 months | At 6 months
  Interval between the date of inclusion in the trial until the date of recurrence of irradiated site (first recurrence, in case of multiple irradiation). Patients that are alive without recurrence at the end of the tiral will be censored
Percentage of Recurrence free survival at 12 months | at 12 months
  Interval between the date of inclusion in the trial until the date of recurrence of irradiated site (first recurrence, in case of multiple irradiation). Patients that are alive without recurrence at the end of the tiral will be censored
Overall survival | From date of inclusion until the date of death from any cause, assessed up to 72 months
  Interval between the date of inclusion in the trial until the date of death whatever the cause. Patients that are alive without recurrence at the end of the tiral will be censored
Tolerance of re-irradiation | up to 24 months
  Recording of toxicities (according to Common Terminology Criteria for Adverse Events v5 criteria) at each follow-up visit
Characterization of PET parameters at recurrence and compare them to baseline parameters with SUV max value | up to 24 months
  Standardized Uptake Value (SUV) max
Characterization of PET parameters at recurrence and compare them to baseline parameters with SUV mean value | up to 24 months
  SUV mean
Characterization of PET parameters at recurrence and compare them to baseline parameters with SUV peak value | up to 24 months
  SUV peak
Quality of Life at 2 months measured with Quality of Life Questionnaire-Cancer 30items (QLQ-C30) | At 2 months
  Quality of life will be measure with the Quality of Life Questionnaire-C30 (Cancer 30items).
  All items are scored 1 (worse outcome) to 4 (better outcome) or 1 (worse outcome) to 7 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life at 2 months measured with Quality of Life Questionnaire-Brain Neoplasms 20items (QLQ-BN20) | At 2 months
  Quality of life will be measured with Quality of Life Questionnaire - BN20 (Brain Neoplasms 20items).
  All items are scored 1 (worse outcome) to 4 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life at 4 months measured with Quality of Life Questionnaire-Cancer 30items (QLQ-C30) | At 4 months
  Quality of life will be measure with the Quality of Life Questionnaire-C30 (Cancer 30items).
  All items are scored 1 (worse outcome) to 4 (better outcome) or 1 (worse outcome) to 7 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life at 4 months measured with Quality of Life Questionnaire-Brain Neoplasms 20items (QLQ-BN20) | At 4 months
  Quality of life will be measured with Quality of Life Questionnaire - BN20 (Brain Neoplasms 20items).
  All items are scored 1 (worse outcome) to 4 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life at 6 months measured with Quality of Life Questionnaire-Cancer 30items (QLQ-C30) | At 6 months
  Quality of life will be measure with the Quality of Life Questionnaire-C30 (Cancer 30items).
  All items are scored 1 (worse outcome) to 4 (better outcome) or 1 (worse outcome) to 7 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life at 6 months measured with Quality of Life Questionnaire-Brain Neoplasms 20items (QLQ-BN20) | At 6 months
  Quality of life will be measured with Quality of Life Questionnaire - BN20 (Brain Neoplasms 20items).
  All items are scored 1 (worse outcome) to 4 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life at 12 months measured with Quality of Life Questionnaire-Cancer 30items (QLQ-C30) | At 12 months
  Quality of life will be measure with the Quality of Life Questionnaire-C30 (Cancer 30items).
  All items are scored 1 (worse outcome) to 4 (better outcome) or 1 (worse outcome) to 7 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Quality of Life at 12 months measured with Quality of Life Questionnaire-Brain Neoplasms 20items (QLQ-BN20) | At 12 months
  Quality of life will be measured with Quality of Life Questionnaire - BN20 (Brain Neoplasms 20items).
  All items are scored 1 (worse outcome) to 4 (better outcome). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU de Nancy, Nancy, De
  - Centre Paul Strauss, Strasbourg